CLINICAL TRIAL: NCT06595342
Title: A Prospective Cohort of Patients With Cervical/Intracranial Arteries Stenosis in China
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yi Yang, The associate deam, The First Hospital of Jilin University
Other Study IDs: ARTERIES
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cervical Artery Stenosis; Intracranial Artery Stenosis
Keywords: Cervical Artery Stenosis; Intracranial Artery Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cervical/intracranial arteries stenosis: Investigators plan to enroll 60000 patients with cervical/intracranial arteries stenosis including mild stenosis, moderate stenosis, severe stenosis or occlusion.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The aim of this study is to establish a prospective cohort of patients with cervical/intracranial arteries stenosis in China.

DETAILED DESCRIPTION:
A prospective cohort of patients with cervical/intracranial arteries stenosis from various regions of China will be established. This prospective cohort is used to identify the distribution of risk factors in the patients with cervical/intracranial arteries stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 and ≤ 80 years;
2. Ultrasound or imaging examinations indicating cervical artery stenosis and/or intracranial artery stenosis (including mild, moderate, severe stenosis, or occlusion);
3. Willing to participate and signing the informed consent form.

Exclusion Criteria:

1. Patients with stroke occurring within the past year;
2. Patients with severe systemic diseases, such as respiratory failure, renal failure, gastrointestinal bleeding, coagulation disorders, malignancies, etc.;
3. Patients with a life expectancy of less than one year or those who are unable to complete the study for other reasons.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with cervical artery stenosis and/or intracranial artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke | One year
  Incidence of stroke events including ischemic stroke, transient ischaemic attack and haemorrhagic stroke.

SECONDARY OUTCOMES:
Changes in the stenosis rate of cervical and intracranial arteries | One year
  The changes in the stenosis rate of cervical and intracranial arteries.
Incidence of new clinical vascular events | One year
  Incidence of new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ transient ischemic stroke/ myocardial infarction/ vascular death) as a cluster and evaluated individually. Vascular death was defined as death due to stroke (ischemic or hemorrhagic), systemic hemorrhage, myocardial infarction, congestive heart failure, pulmonary embolism, sudden death, or arrhythmia.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided